CLINICAL TRIAL: NCT04915989
Title: A Phase 1, Multicenter, Open-Label, Single Arm Study to Investigate the Safety and Immunogenicity of GX-19N, a COVID-19 Preventive DNA Vaccine in Elderly Individuals
Brief Title: Safety and Immunogenicity of GX-19N, a COVID-19 Preventive DNA Vaccine in Elderly Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GX-19N-HV-003
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — GX-19N vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GX-19N (Experimental): Dose A of GX-19N will be intramuscularly administered via Electroporator(EP) on day 1 and day 29. (Optional administration on day 57)
  Interventions: Drug: GX-19N

INTERVENTIONS:
Drug: GX-19N — DNA vaccine expressing SARS-CoV-2 S-protein antigen including the Nucleocapsid protein (NP) antigen
  Other Names: Dose A

SUMMARY:
The objective of the study is to demonstrate safety and immunogenicity of COVID-19 preventive DNA vaccine in elderly individuals.

DETAILED DESCRIPTION:
This clinical study is a phase 1 clinical trial to investigate the safety and immunogenicity of COVID-19 preventive vaccine by intramuscularly administration in the elderly.

This study is designed as single arm, open-labeled and a total of 30 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with all study procedures and voluntarily signs informed consent form
* Male or female aged 55-85 years
* Willing to provide specimens such as blood and urine during the study, including end of study visit.

Exclusion Criteria:

* Immunosuppression including immunodeficiency disease or family history Any history of malignant disease within the past 5 years
* Scheduled to undergo any surgery or dental treatment during the study
* Having received immunoglobulin or blood-derived drugs or being expected to be administered within 3 months prior to administration.
* Having relied on antipsychotic drugs and narcotic analgesics within 6 months before administration
* Positive of serology test at screening
* Suspected of drug abuse or a history within 12 months prior to administration
* Active alcohol use or history of alcohol abuse
* Serious adverse reaction to a drug containing GX-19N or other ingredients of the same categories or to a vaccine or antibiotic, nonsteroidal anti-inflammatory disease control, etc. or an allergic history
* History of hypersensitivity to vaccination such as Guillain-Barre syndrome
* Those with significant chronic underlying diseases that may increase the risk of COVID-19 or interfere with the evaluation of clinical trial purposes according to the investigator's discretion
* Having hemophilia at risk of causing serious bleeding when injected intramuscularly or receiving anticoagulants
* Subjects who have been contact with COVID-19 infections in the past prior to administration, have been classified as COVID-19 confirmed patients, medical patients or patients with symptoms or have been identified with SARS and MERS infection history in the past
* Acute fever, cough, difficulty breathing, chills, muscle aches, headache, sore throat, loss of smell, or loss of taste within 72 hours prior to administration
* Other vaccination history within 28 days prior to the administration or being scheduled to be inoculated during the study
* History of having taken immunosuppressant or Immune modifying drug within 3 months prior to administration
* Having participated and had clinical trial drug administration in another clinical trial or biological equivalence study within 6 months prior to the administration
* Pregnant or breastfeeding female, however, those are allowed to participate in the study only if they stop breastfeeding before participation (fertile female† must be negative in serum pregnancy test at screening
* Fertile female who do not agree to use effective contraception methods (condoms, contraceptive diaphragm, intrauterine contraceptive devices) during the study
* Any other clinically significant medical or psychiatric finding which is considered inappropriate by investigator

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Solicited Adverse Event(AE)s | Through 1 year post vaccination
  solicited local and systemic AEs after vaccination
Incidence of Unsolicited Adverse Events | Through 1 year post vaccination
  unsolicited AEs after vaccination
Incidence of Serious Adverse Event(SAE)s | Through 1 year post vaccination
  percentage of subjects with SAEs

SECONDARY OUTCOMES:
GMT of Antigen-specific Binding Antibody Titers | Through 12 weeks after vaccination
  Geometric mean titer (GMT) of antigen-specific binding antibody after vaccination
GMFR of Antigen-specific Binding Antibody Titers | Through 12 weeks after vaccination
  Geometric mean fold rise (GMFR) of antigen-specific binding antibody after vaccination
Percentage of Subjects Who Seroconverted After Vaccination | Through 12 weeks after vaccination
  Seroconversion defines as 4-fold increase in antibody titer after vaccination
GMT of Neutralizing Antibody Level | Through 12 weeks after vaccination
  Geometric mean titer (GMT) of neutralizing antibody after vaccination
GMFR of Neutralizing Antibody Level | Through 12 weeks after vaccination
  Geometric mean fold rise (GMFR) of neutralizing antibody after vaccination
GMSN of Spot Forming Unit (SFU) detected by interferon(IFN)-gamma ELISPOT assay | Through 12 weeks after vaccination
  Geometric mean spot numbers (GMSN) of SFU after vaccination
GMFR of Spot Forming Unit (SFU) detected by IFN-gamma ELISPOT assay | Through 12 weeks after vaccination
  Geometric mean fold rise (GMFR) of SFU after vaccination

OTHER OUTCOMES:
Change From Baseline in Antigen-specific IFN-gamma Cellular Immune Response by Immunophenotyping assay | Through 12 weeks after vaccination
  Antigen-specific IFN-γ T cell immune response assessed by immunophenotyping assay after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yong Choi, MD, Principal Investigator — Severance Hospital
Locations (2):
- South Korea (2):
  - Severance hospital, Seoul
  - Gangnam Severance hospital, Seoul

IPD SHARING:
Plan to Share IPD: No